CLINICAL TRIAL: NCT00381771
Title: Prevalence of Salivary Hypofunction in Patients With Globus Pharyngeus
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Han-Sin Jeong, Pf, Samsung Medical Center
Other Study IDs: SMC IRB 2006-01-028
Record Dates: First submitted 2006-09-27; First posted 2006-09-28 (Estimated); Last update posted 2010-07-28 (Estimated); Status verified 2010-07

CONDITIONS: Globus Pharyngeus
Keywords: Globus Pharyngeus; Xerostomia; Salivary Hypofunction; Pharyngoxerosis
MeSH Terms: conditions — Globus Sensation; Xerostomia | interventions — Conservative Treatment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Objective salivary function: Based on the salivary scintigraphy,
  1. Objective salivary normo-function
  2. Objective salivary dysfunction
  Interventions: Behavioral: Conservative management for xerostomia

INTERVENTIONS:
Behavioral: Conservative management for xerostomia — Active hydration (drinking more than 10 cups of water per day), Humidification, Oral gargle with a diluted (0.05% to 0.1%) chlorhexidine solution, Sugarless chewing gum, Saliva-stimulating sour juice (sugarless orange juice), Commercial artificial saliva, Nasal saline spray 3 to 4 times a day, Warm massage of the 4 major salivary glands.

SUMMARY:
It is well known that 'globus sensation in throat' is caused by the chronic irritation and inflammation of oral, pharyngeal, or laryngeal mucosa, such as laryngopharyngeal reflux and chronic postnasal drip.

Xerostomia and pharyngoxerosis due to salivary hypofunction also proved to induce the mucosal change of the oral cavity and pharynx.

However, no previous studies have documented the prevalence of salivary hypofunction in patients with globus pharyngeus.

Through this clinical investigation, we hypothesized that the salivary hypofunction might be one of the leading cause of globus pharyngeus.

DETAILED DESCRIPTION:
Subjects: patients with symptoms of globus pharyngeus

Globus symptom scoring: 0(mild) to 5(severe)

Subjective symptom analysis by "Standard Table for Xerostomia and Pharyngoxerosis"

Subjective physical finding analysis by "Standard Table for Xerostomia and Pharyngoxerosis"

Objective analysis of Salivary function by 99m-Tc Salivary scintigraphy

--> Define the prevalence of salivary hypofunction in patients with globus pharyngeus (Primary end point)

Subsequent analysis (Secondary end point)

1. Group 1: Globus patients with objective salivary hypofunction
2. Group 2: Globus patients with normal salivary function

Intervention: Active management for xerostomia (Moisturizing, Gargling, Humidification, Massage of salivary gland, Stimulant of salivary secretion, Artificial saliva)

Evaluation of the change of globus symptoms after active management of xerostomia between the Group 1 and Group 2 (at 1 months, at 3 months after the initiation of intervention)

ELIGIBILITY:
Inclusion Criteria:

* Subjects with globus pharyngeus symptoms

Exclusion Criteria:

* Subjects with tumors in oral cavity, oropharynx, nasopharynx, hypopharynx, which may cause globus symptoms
* subjects, who do not undergo the endoscopic exam for the upper aerodigestive tract including oral cavity, oropharynx, nasopharynx, hypopharynx.
* subjects, who take medications that may have potential effect on the mucosa of the upper aerodigestive tract including oral cavity, oropharynx, nasopharynx, hypopharynx.
* subjects with poor medical performance (<70%)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Globus phryngeus patients (complaining foreign body sensation in the throat, but not having true mass lesions)
Sampling Method: Non-Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2006-02; Primary Completion 2007-08 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Han-Sin Jeong, M.D, Principal Investigator — Samsung Medical Center, Dept of Otorhinolaryngology-Head and Neck Surgery
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea

REFERENCES:
- [Result] Baek CH, Chung MK, Choi JY, So YK, Son YI, Jeong HS. Role of salivary function in patients with globus pharyngeus. Head Neck. 2010 Feb;32(2):244-52. doi: 10.1002/hed.21176. PMID 19572282